CLINICAL TRIAL: NCT00738842
Title: A Randomised, Double-Blind, Two-Period Crossover Study to Assess the Effect of AZD6140 on Uric Acid Levels in Healthy Male Volunteers
Brief Title: Uric Acid Study in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Jay Horrow, MD, Medical Science Director, AZD6140, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D5130C00050
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Gout; Coronary Artery Disease
Keywords: Uric; Acid; Level
MeSH Terms: conditions — Gout; Coronary Artery Disease; Heartburn | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD6140
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo to match AZD6140

INTERVENTIONS:
Drug: AZD6140 — Oral tablets taken bid for 5 days
  Arms: 1
Drug: Placebo to match AZD6140 — Oral tablets taken bid for 5 days
  Arms: 2

SUMMARY:
This study is being conducted to examine the effect of AZD6140 on the levels of certain chemicals in subjects' blood and urine.

ELIGIBILITY:
Inclusion Criteria:

* Normal physical examination, vital signs, electrocardiogram (ECG) and laboratory values (unless the investigator considers an abnormality not to be clinically significant)
* Normal laboratory tests at screening
* Non-smoker (no cigarette/tobacco use for at least 6 months)

Exclusion Criteria:

* Personal or family history of gout, gouty arthritis, or renal stones

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The effect of AZD6140 on the levels of certain chemicals in subjects' blood and urine. | Levels or certain chemicals in subjects' blood and urine will be measured at scheduled times during the first 7 days of the study.

SECONDARY OUTCOMES:
The blood levels of AZD6140 in various subjects on the same diet. | following dosing during the first 5 days of the study
The effect of taking AZD6140 on the levels of certain hormones in urine | during the first 5 days of the study

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — AstraZeneca; Stuart Harris, MD, Principal Investigator — SeaView Research